CLINICAL TRIAL: NCT00605033
Title: A Randomized Acceptability and Safety Study of the Transfer From Subutex to Suboxone in Opioid- Dependent Subjects
Brief Title: A Randomized Acceptability and Safety Study of the Transfer From Subutex to Suboxone in Opioid- Dependent Subjects (Study P04843)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04843; SWITCH
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2010-06-30 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Opiate Dependence; Drug Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suboxone (Active Comparator): Double-blind, once-daily sublingual Suboxone (buprenorphine/naloxone 4 mg/1 mg to 24 mg/6 mg) plus matching Subutex placebo during Week 1 followed by open-label, once-daily sublingual Suboxone (buprenorphine/naloxone 4 mg/1 mg to 24 mg/6 mg) during Weeks 2-4 with weekly access to take-home doses as of Week 2.
  Interventions: Drug: Suboxone, Buprenorphine Hydrochloride + Naloxone, SCH 484
- Subutex (Active Comparator): Double-blind, once-daily sublingual Subutex (buprenorphine 4 mg to 24 mg) plus matching Suboxone placebo during Week 1 followed by open-label, once-daily sublingual Subutex (buprenorphine 4 mg to 24 mg) during Weeks 2-4 with weekly access to take-home doses as of Week 2.
  Interventions: Drug: Subutex, Buprenorphine Hydrochloride, SCH 28444

INTERVENTIONS:
Drug: Suboxone, Buprenorphine Hydrochloride + Naloxone, SCH 484 — Suboxone sublingual tablet 4 mg/1 mg - 24 mg/6 mg, daily for 28 days
  Arms: Suboxone
Drug: Subutex, Buprenorphine Hydrochloride, SCH 28444 — Subutex sublingual tablet 4-24 mg, daily for 28 days
  Arms: Subutex

SUMMARY:
Post-marketing commitment to the European Medicines Agency to conduct a prospective, controlled study of the transfer from Subutex to Suboxone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be males or non-pregnant, non-lactating females.
* Subjects must be at least 15 years of age, of either sex, and any race.
* Subjects (and/or the parent or guardian for subjects under the age of legal consent or who otherwise are unable to provide independent consent) must demonstrate willingness to participate in the study and to adhere to dose and visit schedules.
* Subjects must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria(18) for opioid dependence.
* Subjects must have been receiving maintenance treatment with Subutex at doses ranging from 4 mg to the maximum dose permitted by country labeling requirements, but not to exceed 24 mg/day, for at least 1 month prior to screening.
* Subjects must not, according to self-report, have injected opioids more than four times in the month prior to screening.
* Subjects must have an opioid-negative urine drug screening (UDS) result prior to randomization.
* Each subject must confirm that he or she is practicing adequate contraception.
* Female subjects of childbearing potential must have a negative urine beta-human chorionic gonadotropin (β-hCG) test prior to enrollment in the study.

Exclusion Criteria:

* Subjects for whom treatment with either Subutex or Suboxone as required in the protocol would be inconsistent with national labeling.
* Subjects who are unwilling or unable to comply with the requirements of the protocol (eg, pending incarceration) or are in a situation or condition that, in the opinion of the investigator, may interfere with participation in the study.
* Subjects who are participating in any other clinical study in which medication(s) are being delivered.
* Subjects with known allergy or sensitivity to naloxone.
* Subjects who are on the staff, affiliated with, or a family member of the staff personnel directly involved with this study.
* Subjects must not have serious untreated Axis I DSM-IV-TR psychiatric comorbidity (eg, those who are actively suicidal or homicidal, have untreated schizophrenia, etc). Polysubstance abuse or dependence will not exclude subjects except in the case of unauthorized and significant benzodiazepine use requiring medical detoxification or alcohol dependence requiring medical detoxification.
* Human immunodeficiency virus (HIV)-positive subjects with clinical acquired immunodeficiency syndrome (AIDS).
* Subjects treated with generic buprenorphine.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Suboxone: Double-blind, once-daily sublingual Suboxone (buprenorphine/naloxone 4 mg/1 mg to 24 mg/6 mg) plus matching Subutex placebo during Week 1 followed by open-label, once-daily sublingual Suboxone during Weeks 2-4 with weekly access to take-home doses as of Week 2.
- Subutex: Double-blind, once-daily sublingual Subutex (buprenorphine 4 mg to 24 mg) plus matching Suboxone placebo during Week 1 followed by open-label, once-daily sublingual Subutex during Weeks 2-4 with weekly access to take-home doses as of Week 2.
Period: Overall Study
Arm/Group | Suboxone | Subutex
Started | 143 | 98 (One participant was randomized but withdrew before taking any study medication (treated n=97).)
Completed | 136 | 90
Not Completed | 7 | 8
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suboxone | Subutex | Total
Number analyzed (Participants) | 143 | 97 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (8.2) | 35.5 (8.7) | 35.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 52
  Male | 113 | 75 | 188

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate was defined as the percentage of participants who did not receive a dose increase from the dose given at the first dosing date by Day 7 of a one-week, randomized, double-blind, double-dummy treatment transfer phase.
Time Frame: Assessed by Day 7 of double-blind, double-dummy treatment period.
Population: Analysis of primary outcome was done on the intention-to-treat (ITT) population, defined as all randomized subjects who took at least one dose of study medication and provided at least one valid post-baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Suboxone | Subutex
Number analyzed (Participants) | 143 | 97
Percentage of participants | 83.2 | 88.7
Statistical Analysis 1: Comparison: Suboxone vs Subutex; Test type: Non-Inferiority or Equivalence — Non-inferiority was defined as a lower bound of the two-sided 95% confidence interval of the proportion difference greater than -0.15; Binomial approximation; Proportion difference = -0.054, 95% CI 2-sided [-0.142 to 0.034]

ADVERSE EVENTS:
Arm/Group | Suboxone | Subutex
Serious Adverse Events (participants affected / at risk) | 2/143 | 4/97
Other Adverse Events (participants affected / at risk) | 79/143 | 52/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suboxone (N=143) | Subutex (N=97)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug detoxification (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suboxone (N=143) | Subutex (N=97)
Lacrimation increased (Eye disorders) | 9 (9) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 9 (14) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 21 (29) | 7 (8)
Toothache (Gastrointestinal disorders) | 1 (1) | 5 (5)
Asthenia (General disorders) | 12 (15) | 7 (8)
Chills (General disorders) | 10 (11) | 7 (7)
Fatigue (General disorders) | 7 (8) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 7 (7)
Headache (Nervous system disorders) | 23 (30) | 12 (15)
Anxiety (Psychiatric disorders) | 23 (27) | 16 (17)
Drug dependence (Psychiatric disorders) | 10 (11) | 4 (6)
Restlessness (Psychiatric disorders) | 6 (6) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 6 (6)
Yawning (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 (28) | 9 (11)
Piloerection (Skin and subcutaneous tissue disorders) | 9 (10) | 2 (3)
Hot flush (Vascular disorders) | 10 (12) | 5 (5)
Insomnia (Psychiatric disorders) | 12 (12) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will publish/present results together with other study sites, unless written permission is obtained from Sponsor. Investigator provides 45 days' written notice to Sponsor prior to submission for publication/presentation so that Sponsor can review copies of abstracts/manuscripts reporting results. Sponsor has the right to review/comment on any presentation regarding proprietary information, accuracy and fair balance of the information, and compliance with FDA regulations.